CLINICAL TRIAL: NCT07365904
Title: A Single-centre, Open-label, Phase II Study on the Maintenance of Ovulation Inhibition After Intentional Application Contraceptive
Brief Title: Investigating Ovulation Inhibition for Use as a Contraceptive
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MR-130A-01-TD-2002
Record Dates: First submitted 2025-09-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- "regular": regular application without planned application errors (Experimental)
  Interventions: Drug: MR-130A-01 contraceptive transdermal patch, containing norelgestromin (NGMN)
- Extended Period 1: regular application with planned application errors (Experimental)
  Interventions: Drug: MR-130A-01 contraceptive transdermal patch, containing norelgestromin (NGMN)
- Extended Period 2: regular application with planned application errors (Experimental)
  Interventions: Drug: MR-130A-01 contraceptive transdermal patch, containing norelgestromin (NGMN)

INTERVENTIONS:
Drug: MR-130A-01 contraceptive transdermal patch, containing norelgestromin (NGMN) — MR-130A-01 contraceptive transdermal patch, containing norelgestromin (NGMN)

SUMMARY:
A single-centre, open-label, randomised, phase II study on the maintenance of ovulation inhibition after intentional application errors during 84 days of treatment with MR 130A 01 contraceptive transdermal patch

DETAILED DESCRIPTION:
Ovulation inhibition study of MR-130A-01 contraceptive transdermal patch containing norelgestromin with intentional application errors; MR-130A-01-TD-2002

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy, post-menarcheal and premenopausal women of age 18 to 35 years (inclusive) at screening examination.

  2. BMI ≥18.0 kg/m2 at screening examination. 3. Participants must be in good physical and mental health as determined by vital signs, medical history, and physical and gynecological examination, as assessed by the investigator.

  4. Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the participant participating in the clinical trial.

  5. Status at least 3 months after a delivery, abortion, and stopping lactation, if applicable, before screening.

  6. Has regular menstrual cycles that are between 21 and 35 days in duration as reported by the participant during anamnesis, with an intact uterus and ovaries. If the participant uses hormonal birth control at screening, historic data should be used to evaluate this criterion.

  7. Both ovaries must be visible on TVUS examination during screening. 8. Ovulatory pre-treatment cycle, as confirmed by a progesterone concentration >10.0 nmol/L.

  9. Participants must consent to use reliable non-hormonal contraceptive methods (male condoms, diaphragm, or heterosexual abstinence) throughout the study, unless the participant has a history of female sterilization or sterilization of the sexual partner.

Exclusion Criteria:

* 1. Known hypersensitivity or intolerance to any ingredient of the investigational product.

  2. History or presence of dermal sensitivity to medicated patches or to topical applications including bandages, surgical tape.

  3. Pregnancy or a positive serum beta human chorionic gonadotropin (β-hCG) pregnancy test at screening.

  4. Clinically relevant abnormal findings from serum biochemistry and hematology and HBsAG/ Hepatitis C virus/ human immunodeficiency virus (HIV) serology as evaluated by the investigator 5. ASAT (aspartate-aminotransferase) > 20 % upper limit of normal (ULN), ALAT (alanine-aminotransferase) > 10 % ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL corresponds to > 9 µmol/l ULN).

  6. Use of a non-hormonal intra-uterine device within the pre-treatment cycle or any hormonal contraception as follows:
  * Short-acting hormonal contraceptives such as oral, patch, ring or intrauterine systems within the menstrual cycle prior to the pre-treatment cycle.
  * Injectable (intramuscularly or subcutaneously) within 10 months (three-month treatment duration), 6 months (two-month treatment duration) or 3 months (one-month treatment duration) prior to the start of pre-treatment cycle or implants within the menstrual cycle prior to the pre-treatment cycle.

    7. Known or suspected malignancy or history thereof. 8. Unexplained vaginal bleeding within the past 6 months suspicious for serious condition, or any abnormal bleeding which is expected to recur during the study (e.g. bleeding from cervical polyp, recurrent bleeding after sex).

    9. History or presence of ischemic heart disease, coronary artery disease, myocardial infarction, stroke, other cerebrovascular diseases including transient ischemic attacks (TIAs).

    10. History or presence of hypertension or hypertension with vascular disease or elevated blood pressure (BP) defined as systolic BP ≥140 mm Hg or diastolic BP ≥90 mm Hg, measured in sitting position after at least 5 minutes of rest (a single reading of blood pressure level is not sufficient to classify a woman as hypertensive).

    11. Pulse rate (PR) < 50 bpm or > 90 bpm 12. Presence of deep vein thrombosis/pulmonary embolism. 13. Has any comorbid condition that may require major surgery with prolonged immobilization during the study period.

    14. Presence of liver disease including severe (decompensated) cirrhosis, benign (e.g., hepatocellular adenoma) or malignant liver tumors.

    15. Chronic disease potentially necessitating organ transplantation during the anticipated course of the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Ovulation incidence in cycle with regular application, and in cycles with extended period application errors. Ovulation is defined as a Hoogland-Skouby score 5 or 6 in combination with fulfilment of Landgren criterion. | 84 days

SECONDARY OUTCOMES:
Ovulation incidence overall and incidence per treatment cycle. | 84 days
HSS determined for each treatment cycle. | 84 days
Fulfilment of Landgren criterion in cycles with HSS 5 or 6. | 84 days
FLS diameter and endometrial thickness determined by transvaginal ultrasound (TVUS). | 84 days
Pituitary (luteinizing hormone [LH]) and ovarian (estradiol [E2], progesterone [P]) hormone concentrations in serum. | 84 days
Plasma concentration of NGMN and its metabolite norgestrel Immediately 5min before and at the end of one scheduled patch-free window. | 84 days
Plasma concentrations of NGMN and norgestrel. | 84 days
Assessment of adhesion score by the participants themselves and by the site personnel. | 84 days
Safety and tolerability: Treatment-emergent Adverse Events (TEAE) Safety clinical laboratory parameters Incidence of application site reactions (skin irritation scores assessed by the participants). | 84 days
Bleeding pattern determined as Incidences of bleeding and/or spotting episodes. Number of observed days of bleeding and/or spotting, bleeding only and spotting only. Incidences of complete absence of bleeding or spotting (excluding the first episode). | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jagtap, Study Director — Meda Pharma GmbH & Co. KG (a Viatris company)
Locations (1):
- dinox GmbH, Berlin, Germany